CLINICAL TRIAL: NCT04080336
Title: Comparison of Vaginal Misoprostol and Dinoprostone Prior to Copper Intrauterine Device Insertion in Nulliparous Women:a Randomized Controlled Trial
Brief Title: Comparison of Vaginal Misoprostol and Dinoprostone Prior to Copper Intrauterine Device Insertion in Nulliparous Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: dinoprostone misoprostol IUD
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: IUD Insertion Complication
MeSH Terms: interventions — Dinoprostone; Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dinoprostone (Experimental): 1 vaginal tablet of dinoprostone (3mg) (prostin® E2, Pharmacia & Upjohn, Puurs, Belgium) inserted by the study nurse 3 hours before IUD insertion.
  Interventions: Drug: Dinoprostone
- misoprostol (Active Comparator): 1 vaginal tablet of misoprostol (200 mcg) (Misotac®; Sigma Pharma, SAE, Egypt) inserted by the study nurse 3 hours before IUD insertion.
  Interventions: Drug: Misoprostol
- placebo (Placebo Comparator): one tablet of placebo inserted by the study nurse 3 hours before IUD insertion.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dinoprostone — 1 vaginal tablet of dinoprostone (3mg) (prostin® E2, Pharmacia & Upjohn, Puurs, Belgium) inserted by the study nurse 3hours before IUD insertion.
  Arms: dinoprostone
Drug: Misoprostol — 1 vaginal tablet of misoprostol (200mcg) (Misotac®; Sigma Pharma, SAE, Egypt) inserted by the study nurse 3 hours before IUD insertion.
  Arms: misoprostol
Drug: placebo — one tablet of placebo inserted by the study nurse 3 hours before IUD insertion.
  Arms: placebo

SUMMARY:
To compare the effect of vaginal dinoprostone versus vaginal misoprostol administered before the copper intrauterine device(IUD) insertion in reducing IUD inertion pain and the difficulty in inserting the IUD in nulliparous women.

DETAILED DESCRIPTION:
Long-acting reversible contraception methods are highly effective methods for reduction of the unplanned pregnancy rate worldwide. The intrauterine device is a single procedure that provides reliable, effective and long term contraception for many women. However, the insertion procedure can be associated with a troublesome degree of pain that prevent some women from choosing its use. Different interventions have been described to decrease pain perception during intrauterine device insertion with no agreement on an effective one.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous women requesting copper IUD insertion

Exclusion Criteria:

* pregnancy, Parous women, contraindications or allergy to dinoprostone or misoprostol,contraindication to IUD insertion, untreated active cervicitis or vaginitis, undiagnosed abnormal uterine bleeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
The difference in pain scores during intrauterine device insertion | 10 minutes
  The difference in pain scores during intrauterine device insertion using visual analog scale from 0 to 10

SECONDARY OUTCOMES:
the difference in pain scores during tenaculum application | 10 minutes
  The difference in pain scores during tenaculum application using a visual analog scale from 0 to 10
the difference in pain scores during sound insertion | 10 minutes
  The difference in pain scores during sound insertion using a visual analog scale from 0 to 10
the ease of IUD insertion | 10 minutes
  the ease of IUD insertion using ease of insertion score from 0 to 10 cm (0 = very easy insertion, 10 cm = terribly difficult insertion)
women's satisfaction level | 10 minutes
  women's satisfaction level using satisfaction score from 0 to 10 cm where 0 denotes no satisfaction and 10 denotes maximum satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, Principal Investigator — Cairo University; Mohamed El Sharkawy, Principal Investigator — Cairo University; Mohamed El Mahy, Principal Investigator — Cairo University
Locations (1):
- Ahmed Samy, Giza, Egypt